CLINICAL TRIAL: NCT07374900
Title: Hybrid Versus Fully In-person Physiotherapy for Non-traumatic Shoulder Pain in Routine Care: a Prospective Consecutive Observational Cohort Study
Brief Title: Hybrid Versus Fully In-person Physiotherapy for Non-traumatic Shoulder Pain in Routine Care.
Status: Completed | Type: Observational
Sponsor: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: TDN-REHABI-0120260002; 0011-1408-2022-000012 (Other: Beca de Doctorado Industrial 2022 del Gobierno de Navarra)
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Digital Shoulder Rehabilitation
Keywords: shoulder pain; physiotherapy; hybrid rehabilitation; home exercise; time to discharge; real-world evidence
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 200 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Hybrid rehabilitation: One supervised in-person session plus two remote (non-face-to-face) sessions per week, delivered in 3-week cycles.
- Group 2: In-person rehabilitation: Description:three supervised in-person sessions per week, delivered in 3-week cycles according to the REHABI protocol.

SUMMARY:
Prospective consecutive observational cohort study in routine care comparing hybrid versus fully in-person supervised physiotherapy for non-traumatic shoulder pain/dysfunction delivered under the standardized REHABI program. The primary outcome is time to clinical discharge (days from first visit to discharge). Secondary outcomes include change in pain (VAS/composite VAS) and change in total clinical deficit score from baseline to discharge.

DETAILED DESCRIPTION:
This prospective consecutive observational study was conducted in routine outpatient care at TDN Clínica (Navarra, Spain) to assess whether outcomes differ between two physiotherapy delivery formats for adults with non-traumatic shoulder pain/dysfunction managed under the same standardized digital workflow (REHABI) between March and September 2025. Allocation to format was feasibility-based (non-random) according to routine-care constraints (e.g., work schedule, transport, distance). Both formats were delivered at a nominal frequency of three sessions/week: hybrid (1 supervised in-person session plus 2 unsupervised home sessions supported by smartphone access to prescribed exercises) and fully in-person (3 supervised in-person sessions/week).

REHABI integrates a structured assessment-prescription-reassessment process. Patients completed a standardized 24-test functional battery at baseline (visit 1) and at follow-up evaluations scheduled every 3-5 weeks until clinical discharge. The battery includes measures of strength (digital dynamometry), range of motion (manual goniometry), flexibility, and clinical tests. Pain intensity during test execution was recorded using a 0-10 visual analogue scale (VAS/EVA) in 16 of the 24 tests; a composite VAS was also used to support discharge decisions. Test scoring yields a total clinical deficit score. Clinical discharge was defined within the workflow using explicit criteria (deficit score threshold, symmetric strength, functional ROM, and low pain during tests).

Study objectives: (1) To assess whether time to clinical discharge (days from baseline to discharge) differs between patients managed with hybrid versus fully in-person rehabilitation in routine care. (2) To assess whether changes from baseline to discharge in pain (VAS/EVA and composite VAS, as recorded) and in the total clinical deficit score differ between formats.

ELIGIBILITY:
Inclusion Criteria

* Age 18-71 years
* Non-traumatic shoulder pain/dysfunction
* Access to a smartphone to view exercises
* Completion of a full rehabilitation episode within the study period

Exclusion Criteria:

* Acute fractures or dislocations
* Arthritis/osteoarthritis
* Osteosarcoma or osteomyelitis
* Recent shoulder surgery
* Incomplete rehabilitation episode or missing baseline/discharge data

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with musculoskeletal shoulder pain treated in a private sports physiotherapy clinic in Pamplona, Spain, who are referred or self-referred for conservative management, consecutively enrolled in the REHABI digital rehabilitation program, and who have access to and basic skills to use a smartphone.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Time to clinical discharge | From baseline (V1) until discharge (end of rehabilitation episode, approximately 1 to 6 months after baseline, depending on clinical evolution)
  Days from first visit (baseline, V1) to clinical discharge.

SECONDARY OUTCOMES:
Change in total clinical deficit score | baseline and discharge (approximately 1 to 6 months after baseline, depending on clinical evolution)
  Total deficit score (points) at baseline and discharge; change = baseline - discharge.
Change in pain (VAS / composite VAS) | baseline and discharge (approximately 1 to 6 months after baseline, depending on clinical evolution)
  VAS (0-10) and/or composite VAS at baseline and discharge; change.

CONTACTS AND LOCATIONS:
Overall Officials: José A Sanz, PHD, Study Director — Universidad Pública de Navarra; Igor Setuain, PHD, Study Director — TDN Clinica; Iban Latasa, PHD, Study Director — IED Electronics
Locations (1):
- TDN Clínica Traumatología y Rehabilitación SLP, Noaín, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
At present, there is no plan to share individual participant data (IPD). This is a single-center study with a relatively small sample and detailed clinical assessments, which may increase the risk of re-identification, and the original informed consent did not explicitly cover broad IPD sharing. De-identified summary results will be available in the published manuscript, and additional aggregated information may be considered upon reasonable request.

REFERENCES:
- [Result] Setuain I, Gonzalez-Izal M, Paularena A, Luque JL, Andersen LL, Izquierdo M. A protocol for a new methodological model for work-related shoulder complex injuries: From diagnosis to rehabilitation. BMC Musculoskelet Disord. 2017 Feb 7;18(1):70. doi: 10.1186/s12891-017-1435-2. PMID 28173784